CLINICAL TRIAL: NCT03035981
Title: Assessment of Gastric Emptying and Fullness of Rice With Different Starch Properties
Brief Title: Gastric Emptying of Rice With Different Starch Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1405014904
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior | interventions — fructooligosaccharide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- White rice, low amylose (Experimental): Cooked white rice with low amylose content
  Interventions: Other: White rice, low amylose
- White rice, high amylose (Experimental): Cooked white rice with high amylose content
  Interventions: Other: White rice, high amylose
- White rice, slow (Experimental): Cooked white rice with slow digesting starch
  Interventions: Other: White rice, slow
- White rice, resistant (Experimental): Cooked white rice with resistant starch
  Interventions: Other: White rice, resistant
- Brown rice, low amylose (Experimental): Cooked brown rice with low amylose content
  Interventions: Other: Brown rice, low amylose
- Brown rice, high amylose (Experimental): Cooked brown rice with high amylose content
  Interventions: Other: Brown rice, high amylose
- Fructooligosaccharide (FOS) (Experimental): Fermentable carbohydrate solution
  Interventions: Other: Fructooligosaccharide (FOS)

INTERVENTIONS:
Other: White rice, low amylose — White and brown rice were tested for differences in gastric emptying rate and appetitive response
  Arms: White rice, low amylose
Other: White rice, high amylose — White and brown rice were tested for differences in gastric emptying rate and appetitive response
  Arms: White rice, high amylose
Other: White rice, slow — White and brown rice were tested for differences in gastric emptying rate and appetitive response
  Arms: White rice, slow
Other: White rice, resistant — White and brown rice were tested for differences in gastric emptying rate and appetitive response
  Arms: White rice, resistant
Other: Brown rice, low amylose — White and brown rice were tested for differences in gastric emptying rate and appetitive response
  Arms: Brown rice, low amylose
Other: Brown rice, high amylose — White and brown rice were tested for differences in gastric emptying rate and appetitive response
  Arms: Brown rice, high amylose
Other: Fructooligosaccharide (FOS) — White and brown rice were tested for differences in gastric emptying rate and appetitive response
  Arms: Fructooligosaccharide (FOS)

SUMMARY:
Glycemic carbohydrates are associated with metabolic disturbances, such as type II diabetes, due to rapid digestion of starch into glucose. The specific properties of starch within these foods has been studied for the purpose of slowing their digestion rate and improving related physiological outcomes, such as gastric emptying rate. The current study investigated the relationship among starch digestion, gastric emptying rate and satiety in white and brown rice.

DETAILED DESCRIPTION:
Studies have indicated that starch-based foods with somewhat high amylose content have slower in vitro starch digestion rates, which relate to a low glycemic response. Low glycemic response is associated with delayed gastric emptying rate as well. Therefore, we hypothesized that rice with a slow starch digesting property would delay gastric emptying. White and brown rice with varying amylose contents were used in this study. A 13C-labeled octanoic acid breath test method was used to measure gastric emptying rate, and questionnaires were used to assess hunger and fullness during the testing sessions. Twelve healthy volunteers were recruited to participate in a crossover design study with six rice treatments and outcome measurements were gastric emptying and satiety assessments. One fermentable carbohydrate (fructooligosaccharide, FOS) solution was used to validate the production of breath hydrogen.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index (18 kg/m2 ≤ BMI ≤ 25 kg/m2)

Exclusion Criteria:

* Under any medication
* History of any gastrointestinal disease or surgery
* Diabetes
* Smoker

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | Acute study, 4 hours after consumption of test food
  Breath test was performed using 13C-octanoic acid mixed into test meals
Appetitive response | Acute study, 4 hours after consumption of test food
  Fullness and hunger questionnaire was given at various time points after consumption of test foods

SECONDARY OUTCOMES:
Breath hydrogen | Acute study, 4 hours after consumption of test food
  Hydrogen breath test was performed following ingestion of test meals

IPD SHARING:
Plan to Share IPD: No